CLINICAL TRIAL: NCT06115967
Title: A Phase I, Randomised, Double-blind, Placebo-controlled, Single Ascending Dose Study of Safety, Tolerability, Pharmacokinetics, Pharmacodynamics of Subcutaneous AZD6912 in Healthy Participants
Brief Title: A Study to Assess the Safety, Tolerability, Pharmacokinetics, Pharmacodynamics of Subcutaneous AZD6912 in Healthy Participants
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: AstraZeneca (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Sequential | Masking: Triple | Purpose: Treatment
Other Study IDs: D7130C00001
Record Dates: First submitted 2023-10-16; First posted 2023-11-03 (Actual); Last update posted 2025-12-01 (Actual); Status verified 2025-11

CONDITIONS: Rheumatoid Arthritis
Keywords: Complement factor B; Small interfering ribonucleic acid; CFB messenger ribonucleic acid
MeSH Terms: conditions — Arthritis, Rheumatoid

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (9):
- AZD6912 Dose 1 (Experimental): Participants will receive AZD6912 Dose 1.
  Interventions: Drug: AZD6912
- AZD6912 Dose 2 (Experimental): Participants will receive AZD6912 Dose 2.
  Interventions: Drug: AZD6912
- AZD6912 Dose 3 (Experimental): Participants will receive AZD6912 Dose 3.
  Interventions: Drug: AZD6912
- AZD6912 Dose 4 (Experimental): Participants will receive AZD6912 Dose 4.
  Interventions: Drug: AZD6912
- AZD6912 Dose 5 (Experimental): Participants will receive AZD6912 Dose 5.
  Interventions: Drug: AZD6912
- AZD6912 Dose 6 (Experimental): Participants will receive AZD6912 Dose 6.
  Interventions: Drug: AZD6912
- Placebo (Placebo Comparator): Participants will receive Placebo.
  Interventions: Drug: Placebo
- AZD6912 additional Japanese cohort 1 (Experimental): Participants will receive AZD6912.
  Interventions: Drug: AZD6912
- AZD6912 additional Japanese cohort 2 (Experimental): Participants will receive AZD6912.
  Interventions: Drug: AZD6912

INTERVENTIONS:
Drug: AZD6912 — AZD6912 will be administered as a single sub-cutaneous dose.
  Arms: AZD6912 Dose 1; AZD6912 Dose 2; AZD6912 Dose 3; AZD6912 Dose 4; AZD6912 Dose 5; AZD6912 Dose 6; AZD6912 additional Japanese cohort 1; AZD6912 additional Japanese cohort 2
Drug: Placebo — Placebo will be administered as a single sub-cutaneous dose.
  Arms: Placebo

SUMMARY:
This study will evaluate the safety, tolerability, pharmacokinetics (PK), and pharmacodynamics (PD) of single ascending doses of AZD6912 administered subcutaneously (SC) in healthy participants.

DETAILED DESCRIPTION:
In this First-In-Human (FiH) study, eligible participants will be randomly assigned to 6 cohorts in a 3:1 ratio to receive either a single dose of AZD6912 SC or placebo. The first 2 participants in each cohort will be dosed as a sentinel pair, with one receiving AZD6912 SC and the other receiving placebo.

The study will comprise of, a screening period of 70 days, a treatment period where participants will stay at the Clinical Unit from the day before study intervention administration until at least 240 hours and will be discharged on Day 11. Outpatient visits would start weekly from Day 15, then bi-weekly from Day 43, 4-weekly from Day 99, and 6-weekly from Day 155, with additional follow-up visits approximately every 4 weeks as needed until complement activity returns to the normal range.

The study will last approximately 25 months, including the optional Japanese cohorts, with each participant participating for about 38 weeks or longer until complement activity returns to normal range (per local laboratory).

ELIGIBILITY:
Inclusion Criteria:

* Females must have a negative pregnancy test.
* Contraceptive use by males and females should be consistent with local regulations.
* Have a body mass index (BMI) between 18 and 30 kg/m2 inclusive and weigh at least 50 kg.
* For optional Japanese participants only:

  * Participants must be of Japanese descent defined as: first generation (born to 2 Japanese parents and 4 Japanese grandparents).
  * Born in Japan, and not have lived outside Japan for more than 5 years.
  * Lifestyle, including diet, must not have significantly changed since leaving Japan.

Exclusion Criteria:

* History of any clinically important disease or disorder.
* Current or recurrent disease of clinical significance that could affect clinical assessments or clinical laboratory evaluations.
* Any clinically important illness, medical/surgical procedure or trauma within 4 weeks of the first administration of study intervention.
* History of congenital or acquired immunodeficiency or complement deficiency or an underlying condition that predisposes to infection.
* History of any Neisseria infection, unexplained, recurrent infections, or infection requiring treatment with systemic antibiotics.
* Evidence of hepatitis B infection (positive for HBsAg or positive for anti-HBcAb) or hepatitis C viral infection (HCV Abs or hepatitis C RNA positive) or HIV infection (positive for HIV type 1 or type 2 Abs).
* Participants testing positive for COVID-19 prior to dosing.
* Any cardiac abnormalities.
* A CAP activity < 60% at screening.
* Known or suspected history of drug abuse, history of alcohol abuse or smoking.

Ages: 18 Years to 50 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 40 (Actual)
Dates: Start 2023-11-15 (Actual); Primary Completion 2025-10-16 (Actual); Study Completion 2025-10-16 (Actual)

PRIMARY OUTCOMES:
Number of participants with adverse events (AEs) | From screening (Day -70) to last follow up visit (Day 197- approximately 38 weeks)
  To assess the safety and tolerability of AZD6912 in healthy participants.

SECONDARY OUTCOMES:
Maximum observed plasma (peak) drug concentration (Cmax) of AZD6912 | From randomization to Day 197 (up to 28 weeks)
  To characterise the Cmax of single ascending doses of AZD6912 in healthy participants.
Area under plasma concentration-time curve from zero to infinity (AUCinf) of AZD6912 | From randomization to Day 197 (up to 28 weeks)
  To characterise AUCinf of single ascending doses of AZD6912 in healthy participants.
Area under the plasma concentration-curve from zero to the last quantifiable concentration (AUClast) of AZD6912 | From randomization to Day 197 (up to 28 weeks)
  To characterise the AUClast of single ascending doses of AZD6912 in healthy participants.
Time to reach peak or maximum observed concentration or response following drug administration (tmax) of AZD6912 | From randomization to Day 197 (up to 28 weeks)
  To characterise tmax of single ascending doses of AZD6912 in healthy participants.
Time of last measurable concentration (tlast) of AZD6912 | From randomization to Day 197 (up to 28 weeks)
  To characterise tlast of single ascending doses of AZD6912 in healthy participants.
Terminal elimination half-life (t½λz) of AZD6912 | From randomization to Day 197 (up to 28 weeks)
  To characterise t½λz of single ascending doses of AZD6912 in healthy participants.
Dose normalised AUClast (AUClast/D) of AZD6912 | From randomization to Day 197 (up to 28 weeks)
  To characterise AUClast/D of single ascending doses of AZD6912 in healthy participants.
Dose normalised AUCinf (AUCinf/D) of AZD6912 | From randomization to Day 197 (up to 28 weeks)
  To characterise AUCinf/D of single ascending doses of AZD6912 in healthy participants.
Dose normalised Cmax (Cmax/D) of AZD6912 | From randomization to Day 197 (up to 28 weeks)
  To characterise Cmax/D of single ascending doses of AZD6912 in healthy participants.
Apparent total body clearance of drug from plasma after extravascular administration (CL/F) of AZD6912 | From randomization to Day 197 (up to 28 weeks)
  To characterise CL/F of single ascending doses of AZD6912 in healthy participants.
Volume of distribution (apparent) at steady state following extravascular administration (based on terminal phase) (Vz/F) of AZD6912 | From randomization to Day 197 (up to 28 weeks)
  To characterise Vz/F of single ascending doses of AZD6912 in healthy participants.
Percent change from baseline in plasma concentrations of Complement factor B (CFB) protein | From randomization to Day 197 (up to 28 weeks)
  To assess the PD effects of single ascending doses of AZD6912 in healthy participants.
Percent change from baseline in serum of Complement functional activity (CAP) | From randomization to Day 197 (up to 28 weeks)
  To assess the PD effects of single ascending doses of AZD6912 in healthy participants.

CONTACTS AND LOCATIONS:
Locations (2):
- Research Site, Montreal, Quebec, Canada
- Research Site, Harrow, United Kingdom

IPD SHARING:
Plan to Share IPD: Yes
Qualified researchers can request access to anonymized individual patient-level data from AstraZeneca group of companies sponsored clinical trials via the request portal Vivli.org. All requests will be evaluated as per the AZ disclosure commitment: https://astrazenecagrouptrials.pharmacm.com/ST/Submission/Disclosure. "Yes", indicates that AZ are accepting requests for IPD, but this does not mean all requests will be approved.
Supporting Information: Study Protocol
Time Frame: AstraZeneca will meet or exceed data availability as per the commitments made to the EFPIA/PhRMA Data-Sharing Principles. For details of our timelines, please refer to our disclosure commitment at https://astrazenecagrouptrials.pharmacm.com/ST/Submission/Disclosure.
Access Criteria: When a request has been approved AstraZeneca will provide access to the anonymized individual patient-level data via secure research environment Vivli.org. A Signed Data Usage Agreement (non-negotiable contract for data accessors) must be in place before accessing requested information.
URL: https://astrazenecagroup-dt.pharmacm.com/DT/Home